CLINICAL TRIAL: NCT06444568
Title: Efficacy of Modified Ketogenic Diet in Amnestic Mild Cognitive Impairments
Brief Title: Modified Ketogenic Diet in Amnestic Mild Cognitive Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Mehmet Ilkin Naharci, Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKD001
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-06

CONDITIONS: Amnestic Mild Cognitive Disorder; Amnestic Mild Cognitive Impairment
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive control group (No Intervention): The passive control arm will not receive any intervention and will only be evaluated for primary outcome variables at the beginning (week: 0) and at the end (week: 12) of the protocol.
- Active control group (Active Comparator): MIND diet will be applied to participants assigned to the active control arm for 12 weeks. This group will be evaluated at visits (week: 0-4-8-12) in terms of primary and secondary outcome variables, in parallel with the intervention group (KD).
  Interventions: Other: Dietary Intervention
- Intervention group (Modified ketogenic diet) (Experimental): The modified ketogenic diet (MKD) will be applied to participants assigned to the intervention arm for 12 weeks. This group will be evaluated for primary and secondary outcome variables at visits (weeks 0-4-8-12).
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — The intervention includes the application and follow-up of different diet therapies to individuals (Ketogenic diet and MIND).
  Arms: Active control group; Intervention group (Modified ketogenic diet)

SUMMARY:
This clinical study aims to examine the effectiveness of a 12-week modified ketogenic diet (MKD) intervention, especially on cognitive functions, in individuals diagnosed with amnestic-mild cognitive impairment (aMCI) and to compare the effects of control groups (passive or active).

Accordingly, a sample of 36 older adults aged 65-80 years diagnosed with aMCI will be randomized into 3 different groups: passive control (without any intervention), active control (MIND: Mediterranean-DASH Intervention for Neurodegenerative Delay diet) or intervention (MKD). They will be monitored according to targeted criteria throughout the 12-week study protocol.

The main questions this study aims to answer are:

* Does a 12-week MKD intervention improve cognitive functions in aMCI?
* Does the effectiveness of the 12-week MKD intervention in aMCI (i.e., in terms of cognitive function, physical and functional measures, or metabolic/inflammatory biomarkers) differ from control groups?

Expected from participants during the study protocol:

* Participants assigned to the passive control arm are expected to come to the research center at the beginning (week 0) and end (week 12) of the protocol and participate in evaluations.
* Participants assigned to the active control (MIND diet) or intervention (MKD) arm are expected to adhere to assigned dietary therapy, keep a weekly food diary, and have weekly phone calls or online meetings with the dietitian to follow up on the diet. These participants assigned to the diet groups are expected to come to the research center at weeks 0, 4, 8, and 12 to participate in the evaluations.

DETAILED DESCRIPTION:
This study is an open-label, parallel-group randomized controlled clinical trial. The researchers hypothesized that a 12-week modified ketogenic diet (MKD) intervention in participants diagnosed with amnestic-mild cognitive impairments (aMCI) would improve cognitive functions and progression criteria compared to control groups.

The research sample will consist of individuals diagnosed with aMCI, and 36 volunteers, 12 individuals, were randomly assigned to three different research arms according to the block randomization method. To evaluate this sample size in the "repeated measures ANOVA" test of three independent groups with a medium effect size (f:0.30), 5% significance level (α), and 90% power (1-β) in the power analysis, the sample size should be at least 27 individuals has been calculated.

According to the dropout rate (25%) reported in similar ketogenic diet intervention studies in the literature, 36 was targeted as the sample size of the study.

For confidentiality purposes, the coding method will be used in the processing of data according to the study arms and the order of inclusion in the protocol (i.e., PC-1, AC-1, or KD-1, passive/active control, and the ketogenic diet, respectively). It is planned to evaluate cognitive functions with ADAS-Cog (Alzheimer's Disease Assessment Scale: Cognitive Subscale), physical performance with motor-cognitive dual-task and hand grip strength, and functional capacity with Lawton instrumental activities of daily living scale. Yesavage Geriatric Depression Scale-short form (GDS-15), which will also be used as an eligibility criterion, will be used to evaluate mood.

Intervention: After examining the food consumption diaries (7 days), diet planning will be made for the appropriate study arm (MIND or MKD). The daily energy of the diets is eucaloric in two diet groups, and daily energy will be determined according to the daily average energy intake determined by the nutritional status assessment of the individual and the ESPEN (European Society for Clinical Nutrition and Metabolism) consensus recommendation.

Ketogenic diet calculations will be made through the KetoDietCalculator program. The two basic principles of the planned modified ketogenic diet are 1) protein intake of 1 g/kg per day, and 2) a ketogenic diet ratio 1:1. According to the determined daily energy intake, the contribution of macronutrients to daily energy will be determined by the ketogenic diet ratio. Controlling protein intake per body weight is not a routine practice in ketogenic diet applications, and in this study - to preserve lean body mass as much as possible in elderly individuals - the ESPEN consensus recommendation will be taken into account in the calculations.

The MIND diet, which is the control group diet, will be planned following the 14 dietary guidelines defined elsewhere, and the above criteria will be applied in the same way in determining daily energy. MIND is a diet whose neuroprotective properties are currently accepted, with its ability to delay cognitive function loss and dementia supported by many population-based prospective studies.

Following the dietary training, both groups will be given brochures containing the basic principles and instructions of the diet and educational materials containing recipes developed specifically for the diet group. Compliance with the ketogenic diet is evaluated according to the individuals' serum ketone level (compliance criterion: β-hydroxybutyrate/BHB: 0.5-2.5 mmol/L) and food consumption diaries evaluated at 4, 8, and 12 weeks. Compliance with the MIND diet, which is the active control diet, will be evaluated with the MIND diet score calculated from weekly food consumption diaries (compliance criterion: MIND score >10/14).

In evaluating all outcome variables, the per-protocol analysis method will be applied to examine only participants who completed the research protocol. The intention-to-treat method will be used to evaluate some secondary outcome variables (i.e., biomarkers and anthropometry). Changes in primary and secondary outcome variables between the intervention and control groups during the study will be evaluated by repeated measures ANOVA test. All statistical tests will be evaluated in the SPSS (Statistical Package for Social Science) program at 90% power and 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with "amnestic mild cognitive impairment/disorder (aMCI)" by the clinician after the evaluation of cognitive functions according to the neuropsychological evaluation method (0.5 according to the Clinical Dementia Rating Scale (CDR).)
* Having at least 6 years of education.

Exclusion Criteria:

* Under the age of 65 or over the age of 80.
* Diagnosis of neurological (other than MCI) or psychological diseases.
* GDS-15 score > 5 (baseline)
* Kidney/pancreas/liver diseases or dysfunctions, Type 1 diabetes (and Type II diabetic patients receiving insulin replacement therapy), cancer, metabolic diseases (fatty acid oxidation defect, etc.), thyroid dysfunction, pulmonary or autoimmune diseases, head trauma, history of any cardiovascular event (i.e., stroke, myocardial infarction) in the last year.
* Hypercholesterolemia (fasting T-C >300 mg/dL or LDL-C >200 mg/dL), non-reference B12 or folate levels according to biochemical tests performed in the last year.
* Nutritional risks (chewing/swallowing difficulties, history of involuntary weight loss in the last 6 months, body mass index < 22 kg/m2).
* Use of internal device/implant (pacemaker or hearing aid, etc.).
* Medication use (individuals using anticholinergic, antidementia, and opioid class drugs will be excluded; individuals using antidepressant class drugs will be included in the study on the condition that it has been continued for at least 3 months and there is no change in drug type and dose during the study protocol.)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog score | Baseline (week:0) - end of the protocol (week:12)
  Cognitive functions will be evaluated with the ADAS-Cog (Alzheimer's Disease Assessment Scale: Cognitive Subscale) test. This widely used test to assess global cognition, evaluates memory, language, praxis, and orientation with scores ranging from 0 (minimum) to 70 (maximum); increasing scores indicate poorer cognitive performance.

SECONDARY OUTCOMES:
Dual-task (Physical performance) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  Motor-cognitive dual-task testing will be administered to evaluate physical performance. The determined motor and cognitive tasks are 4 meters walking speed and counting backward from 20, respectively, and time (seconds) will be recorded during these tasks. (baseline and end of the protocol for passive control, all visits for active control or intervention groups).
Handgrip strength (kg) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  Hand grip strength will be recorded to evaluate physical performance. The measurement will be performed using the Takei T.K.K.5401 Grip-D digital hand dynamometer (Takei Scientific Instruments Co., Ltd, Japan) and will be repeated twice with both hands and the average score (kg) will be recorded. (baseline and end of the protocol for passive control, all visits for active control or intervention groups).
Total cholesterol (TC, mg/dL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of total cholesterol (TC, mg/dL) was planned to evaluate the effect of dietary intervention on the lipid profile.
Low-density lipoprotein cholesterol (LDL-C, mg/dL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of low-density lipoprotein cholesterol (LDL-C, mg/dL) was planned to evaluate the effect of dietary intervention on the lipid profile.
High-density lipoprotein cholesterol (HDL-C, mg/dL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of high-density lipoprotein cholesterol (HDL-C, mg/dL) was planned to evaluate the effect of dietary intervention on the lipid profile.
Tumor Necrosis Factor-alpha (TNF-α, pg/mL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of Tumor Necrosis Factor-α (TNF-α) was planned to evaluate the effect of dietary intervention on the inflammatory response.
β-hydroxybutyrate (β-HB, mmol/L) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  Within the scope of the research, serum β-HB was planned at all the visits to monitor compliance with the ketogenic diet. (compliance criteria: β-HB: 0,5-2,5 mmol/L).
Serum malondialdehyde (MDA) (nmol/mL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of serum malondialdehyde (MDA) was planned to evaluate the effect of dietary intervention on lipid peroxidation.
Serum Glutathione peroxidase (GSH-Px, U/mL) | Baseline (week:0) - end of the protocol (week:12)
  Within the scope of the research, the measurement of serum Glutathione Peroxidase (GSH-Px) activity was planned to evaluate the effect of dietary intervention on oxidative state.

OTHER OUTCOMES:
Geriatric Depression Scale-short form (GDS-15) score | Baseline (week:0) - end of the protocol (week:12)
  GDS-15 scores will be evaluated to assess mood at the baseline and end of the protocol visits. This scale evaluates mood between 0 (minimum) and 15 (maximum) scores; scores of 0-4 are considered normal, 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Body weight (kg) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  The body weight (kg) will be measured with a Tanita SC330 body composition analyzer (Tanita Health Co., Ltd., Tokyo, Japan) at planned visits throughout the protocol (baseline and end of the protocol for passive control, all visits for active control or intervention groups).
Body height (cm) | Baseline (week:0)
  The height assessment will be performed using a SECA 220 stadiometer (Seca Ltd., United Kingdom) fixed to the wall and recorded in cm.
Body Mass Index (BMI, kg/m^2) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  The body mass index (BMI) will be calculated by dividing the measured body weight (kg) by the square of the height (m). The BMI will be calculated and recorded throughout the protocol (baseline and end of the protocol for passive control, all visits for active control or intervention groups).
Fat-free mass (kg, via body composition analysis) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  Body composition will be analyzed via bioelectrical impedance analysis (BIA) using a Tanita SC330 body composition analyzer (Tanita Health Co., Ltd., Tokyo, Japan). The fat-free mass (kg) obtained as a result of this analysis will be recorded to examine the effects of the intervention at visits planned throughout the protocol. (baseline and end of protocol for passive control, all visits for active control or intervention groups).
Fat mass (kg, via body composition analysis) | Baseline (week:0) - week:4 - week:8 - end of the protocol (week:12)
  Body composition will be analyzed via bioelectrical impedance analysis (BIA) using a Tanita SC330 body composition analyzer (Tanita Health Co., Ltd., Tokyo, Japan). The fat mass (kg) obtained as a result of this analysis will be recorded to examine the effects of the intervention at visits planned throughout the protocol. (baseline and end of protocol for passive control, all visits for active control or intervention groups).
Weekly reported side effects relevant ketogenic diet | week 0-12
  Reported side effects will be recorded weekly only in the MKD arm to monitor compliance and tolerance to the ketogenic diet.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet I Naharcı, Prof., Study Chair — Saglik Bilimleri University
Locations (1):
- Gulhane Faculty of Medicine & Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neth BJ, Mintz A, Whitlow C, Jung Y, Solingapuram Sai K, Register TC, Kellar D, Lockhart SN, Hoscheidt S, Maldjian J, Heslegrave AJ, Blennow K, Cunnane SC, Castellano CA, Zetterberg H, Craft S. Modified ketogenic diet is associated with improved cerebrospinal fluid biomarker profile, cerebral perfusion, and cerebral ketone body uptake in older adults at risk for Alzheimer's disease: a pilot study. Neurobiol Aging. 2020 Feb;86:54-63. doi: 10.1016/j.neurobiolaging.2019.09.015. Epub 2019 Sep 26. PMID 31757576
- [Background] Phillips MCL, Deprez LM, Mortimer GMN, Murtagh DKJ, McCoy S, Mylchreest R, Gilbertson LJ, Clark KM, Simpson PV, McManus EJ, Oh JE, Yadavaraj S, King VM, Pillai A, Romero-Ferrando B, Brinkhuis M, Copeland BM, Samad S, Liao S, Schepel JAC. Randomized crossover trial of a modified ketogenic diet in Alzheimer's disease. Alzheimers Res Ther. 2021 Feb 23;13(1):51. doi: 10.1186/s13195-021-00783-x. PMID 33622392
- [Background] Liu X, Morris MC, Dhana K, Ventrelle J, Johnson K, Bishop L, Hollings CS, Boulin A, Laranjo N, Stubbs BJ, Reilly X, Carey VJ, Wang Y, Furtado JD, Marcovina SM, Tangney C, Aggarwal NT, Arfanakis K, Sacks FM, Barnes LL. Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) study: Rationale, design and baseline characteristics of a randomized control trial of the MIND diet on cognitive decline. Contemp Clin Trials. 2021 Mar;102:106270. doi: 10.1016/j.cct.2021.106270. Epub 2021 Jan 9. PMID 33434704
- [Background] de Crom TOE, Mooldijk SS, Ikram MK, Ikram MA, Voortman T. MIND diet and the risk of dementia: a population-based study. Alzheimers Res Ther. 2022 Jan 12;14(1):8. doi: 10.1186/s13195-022-00957-1. PMID 35022067
- [Background] Kheirouri S, Alizadeh M. MIND diet and cognitive performance in older adults: a systematic review. Crit Rev Food Sci Nutr. 2022;62(29):8059-8077. doi: 10.1080/10408398.2021.1925220. Epub 2021 May 14. PMID 33989093